CLINICAL TRIAL: NCT04555642
Title: Early Diagnosis of Therapy-associated Cardiotoxicity Basing on Multi-tracer Multimodality PET/MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Xuejuan Wang,MD, Principal Investigator, Peking University Cancer Hospital & Institute
Other Study IDs: XW-Heart-001
Record Dates: First submitted 2020-08-31; First posted 2020-09-21 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Positron-Emission Tomography; Magnetic Resonance Imaging
Keywords: Positron-Emission Tomography; cardiotoxicity; Magnetic Resonance Imaging; FDG; FAPI
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- therapy group: lymphoma patients planned chemotherapy or immunotherapy scheme
- healthy control group: Inclusion criteria for the controls were no known diseases or syndromes, within the age range from 18 to 35 years.

SUMMARY:
Using Multi-tracer to early diagnosis of therapy-associated cardiotoxicity using multimodality PET/MRI.

DETAILED DESCRIPTION:
In this study investigators evaluated cardiac uptake by different molecular probe such as FDG, FAPI-04 using multimodality PET/MRI. Previous studies have shown that increased cardiac uptake of FDG on PET may be an indicator of myocardial injury after chemotherapy. Cardiac magnetic resonance (CMR) allows for multiparametric evaluation of cardiac morphology, ventricular function, myocardial perfusion, and viability. The combination of PET with MR (PET/MR) is therefore an alternative attractive pairing for diagnostic imaging. The aim of this study is to find noninvasive and effective method for early diagnosis of cardiotoxicity after chemotherapy or immunotherapy

ELIGIBILITY:
Inclusion Criteria:

* availability of a clinical pre- and post-therapy clinical evaluation encompassing electrocardiogram (ECG) ;
* normal findings at pre-therapy clinical evaluation;
* cancer planned chemotherapy or immunotherapy scheme ;
* available staging FDG-PET/CT scan (PET0);

Exclusion Criteria:

* cannot lie supine for half an hour;
* refuse to join the clinical researcher;
* without metal implants.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with malignant tumor after chemotherapy or immunotherapy
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-12-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
SUVR | 150 days
  the ratio of the standardized uptake value(SUVR) of multi-tracer for the heart within each time window to that of the normal tissue such as hepatic blood pool、blood pool and gluteus.

SECONDARY OUTCOMES:
Change Of Mapping Value and LVEF From Baseline | 150 days
  The change of mapping value and left ventricular ejection fraction between the value before treatment and the value after treatment was calculated based on cardiac magnetic resonance

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Yang, PhD, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No